CLINICAL TRIAL: NCT03553316
Title: A Randomized, Open Labeled, Multiple Dose, 2-Sequence, 2-Period Cross-over Phase 1 Study to Evaluate the Drug-Drug Interaction of PK101-001 and PK101-002 in Healthy Volunteers.
Brief Title: Drug-Drug Interaction Between PK101-001 and PK101-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PMG Pharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK101_P101
Record Dates: First submitted 2018-05-27; First posted 2018-06-12 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2018-08

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence (1) (Experimental): Number of Subject: 24
  Wash out Period: over 7 days (between each period)
  Investigators Products(IPs) for Period1: A (Single)= PK101-002
  IPs for Period2: B (Combination)= PK101-001, PK101-002
  Interventions: Drug: PK101-002; Combination Product: PK101
- Sequence (2) (Experimental): Number of Subject: 24
  Wash out Period: over 7 days (between each period)
  IPs for Period1: B (Combination)= PK101-001, PK101-002
  IPs for Period2: A (Single)= PK101-002
  Interventions: Drug: PK101-002; Combination Product: PK101

INTERVENTIONS:
Drug: PK101-002 — -(Single) PK101-002
  Other Names: A
Combination Product: PK101 — -(Combination) PK101-001, PK101-002
  Other Names: B

SUMMARY:
To evaluate the drug-drug interaction of PK101-001 and PK101-002 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ≥ 19 years of age (on the day of screening)
* No congenital or chronic diseases and no abnormal signs determined by medical examinations
* Not abnormal or not clinical significant lab values
* 90mmHg ≤ (SBP) ≤ 139mmHg, 60mmHg ≤ (DBP) ≤ 89mmHg
* 18Kg/(m)^2 ≤ (BMI) ≤30Kg/(m)^2

Exclusion Criteria:

* Subjects who were administered below medications within 30 days (barbiturates, drugs of induced or suppressive drug metabolizing enzyme, etc)
* Subjects who were administered medications of prohibition within 10 days
* Heavy drinking within 30 days (female: over 14units/week, male:over 21units/week)
* Heavy smoker within 30 days (over 20 cigarettes per day)
* Subjects who previously participated in other clinical trials or bioequivalence Test within 90 days
* Subjects who donated whole blood within 60 days or donated component blood within 14 days or received blood transfusion within 30 days
* Subjects who have hypersensitivity for investigational products

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
AUCτ | 0, 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Area under the plasma drug concentration-time curve for PK101-002 at Steady-state (between dose times)
Cmax,ss | 0, 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  The maximum (or peak) serum concentration for PK101-002 at Steady-state

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hyun Kang, Principal Investigator — H Plus Yangji Clinical Research Center
Locations (1):
- H Plus Yangji Clinical Research Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No